CLINICAL TRIAL: NCT05611138
Title: Växtbaserade Proteiners påverkan på tarmhälsa Hos människa
Brief Title: Dietary Proteins: Metagenomic and Metabolomics Approaches for Human Biomarkers Identification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PanProtein 2
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Healthy male and female adult subjects (n=87) will be recruited to take part in a double-blinded, randomized, 3-arms parallel trial. Subjects that are eligible to take part in the study will be blinded and randomly allocated to consume an isolated plant protein (arm 1) or isolated animal protein (arm 2) or plant-based source of protein (arm 3). The subjects eligible to take part in this study will consume the proteins for 4 weeks, before the intervention they will have a baseline of two weeks, and after the intervention, they will have more two visits. Faecal and blood samples will be used to answer the main outcome of gut-related metabolites and microbiota profile. Blood and urine samples will be used to measure health status and compliance (protein intake markers). Questionnaires will be used to access gastrointestinal symptoms and bowel movement, physical activity level and dietary intake.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isolated pea protein (Experimental): Dietary supplementation with isolated pea protein powder. Amount: 0.5 g of protein from the supplement per kilogram of body weight, taken in 3 portions during the day, for 4 weeks.
  Interventions: Dietary Supplement: Protein supplementation
- Isolated whey protein (Experimental): Dietary supplementation with isolated whey protein. Amount: 0.5 g of protein from the supplement per kilogram of body weight, taken in 3 portions during the day, for 4 weeks.
  Interventions: Dietary Supplement: Protein supplementation
- Concentrated pea protein (Experimental): Dietary supplementation with concentrated pea protein Amount: 0.5 g of protein from the supplement per kilogram of body weight, taken in 3 portions during the day, for 4 weeks.
  Interventions: Dietary Supplement: Protein supplementation

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Participants will be instructed to dissolve the protein powder in liquids (such as water) or on their food (e.g., yoghurt, oat porridge). A subset of the participants (max. 15 per arm) for visits 2 and 6 will be invited to participate in a postprandial challenge, where they will receive the daily protein portion as breakfast.

SUMMARY:
This project aims to create a methodological framework, including the discovery and validation of novel biomarker panels to decipher the impact of plant-based protein intake on health biomarkers. Moreover, the possibility of predicting biomarkers production will be tested by a colonic in vitro fermentation study using study participants' faecal samples.

DETAILED DESCRIPTION:
This study consists of a double-blind, randomised, 3-arm parallel trial, consisting of 2-wk baseline measurements, 4-wk intervention period (with weekly sample collection), and 2-wk after-intervention follow-up, with healthy subjects in each arm consuming different protein sources (from plant- or animal-based sources). Subjects that are eligible to take part in this study will be blinded and randomly allocated to consume an isolated pea protein (arm 1), animal protein (arm 2) or more complex protein pea protein powder (arm 3). The isolated plant and animal protein will be used to evaluate the specific effects of the proteins from the different sources. The more complex protein pea protein powder will be used as a more complex food matrix, containing other food components than protein, to assess how other pea components may impact the specific protein effects. Regardless of the differences in their structure, all supplement powders will be adjusted to provide the same amount of protein. The protein calculation will be done exclusively for each participant, based on their body weight (kg). They will consume up to 2 g of protein per body weight per day. Subjects will be asked to maintain their usual diet and their food intake will be accompanied during the intervention.

Participants' compliance will be followed by their food diaries and by clinical markers for protein intake and will collect blood, faeces and 24 h urine samples. A subset of the participants (max. 15 per arm) for visits 2 and 6 will be invited to participate in a postprandial challenge. After the fastening blood sample collection, they will receive the daily protein portion as breakfast. For those, 9 blood sample time points will be taken, being at 0, 15, 30, 60, 90, 120, 150, 180, and 480 min. After the 180 min measurement, they will receive a standard meal as lunch (e.g., pasta with tomato sauce).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Body mass index (BMI) 18,5-30 kg/m2
* Weight stable within the previous 3 months
* Maintenance of the usual physical activity habits during the study
* Intake of fibre between 15 and 25 g per day (evaluated by 3 food diaries or 24-hours recalls)
* Omnivores

Exclusion Criteria:

* Acute chronic disease, inflammatory or functional gastrointestinal diseases and any other disease or disorder that could affect the outcome of the study
* Use of a medication that may interfere the study outcome
* Eating disorder
* High protein intake (more than 15% of energy or maximum 1,2 g of protein per kg of body weight per day; evaluated by 3 food diaries or 24-hours recalls)
* Use of antibiotic medication during the last 3 months prior the first visit
* Use of antibiotic medication very early in life (e.g., asthmatic children or ear inflammation)
* Use of laxative or anti-diarrhoea medication within the past 3 months before the study
* Regular consumption of probiotic or prebiotic product for the past 6 weeks before the study
* Special diet that is considered to affect the study participation and/or study results, for example, high protein diets
* More than 5 h of moderate-vigorous exercise per week
* Pregnancy or breastfeeding
* Intolerance to dietary supplements that will be used in the study
* Smoking
* Abuse of alcohol or drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Changes in the faecal metabolites using targeted and untargeted metabolomics during the intervention | 8 weeks
  Difference in faecal metabolites depending on the protein supplementation amount and from colonic in vitro fermentation. Targeted and untargeted metabolomics measurements will be used (e.g., short-chain fatty acids and branched chain fatty acids analyses, and polar and non polar metabolomics). Faecal samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared throughout the whole study.
Changes in the plasma metabolites using targete and untargeted metabolomics during the intervention | 4 weeks
  Difference in plasma metabolites (blood obtained fastened state) depending on the protein supplementation amount. Targeted and untargeted metabolomics measurements will be used (e.g., lipids, and polar and non polar metabolomics). Plasma samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared throughout the whole study.
Profile/composition of the gut microbiota during the intervention | 8 weeks
  Difference in the gut microbiota profile/composition because of the protein supplementation and from colonic in vitro fermentation will be assessed by 16s/NGS. Alpha and Beta diversity will be measured and compared throughout the 4 weeks of intervention and baselines. In the case of NGS, the genome sequence will be annotated and the resulting set of genes encoding for metabolic enzymes will be extracted. Data from shotgun metagenomics and metabolomics will be integrated by constructing dependency networks, with a special attempt to infer causal relationships among different variables.
Routinely analysed markers for protein intake/compliance during the intervention - urine | 4 weeks
  Difference in 24 h urine samples markers due to the protein supplementation (e.g., for 24 h urine: urea nitrogen from 24 h urine, creatinine, uric acid)
Routinely analysed markers for protein intake/compliance during the intervention - blood | 4 weeks
  Difference in blood (serum) samples markers due to the protein supplementation (e.g., urea and creatinine)
Changes in the plasma metabolites using targeted and untargeted metabolomics during the dietary challenge | 4 weeks
  Difference in plasma metabolites depending on the protein taken as breaskfast. Targeted and untargeted metabolomics measurements will be used (e.g., polar and non polar metabolomics). Plasma samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared with those found in the fastening state.
Colonic in vitro fermentation | 4 weeks
  Subjects will have their fresh faecal samples used in the colonic in vitro fermentation experiment to evaluate whether and how gut metabolites production can be predicted in vitro. The same proteins used in the dietary intervention study will be digested in vitro and used for the batch in vitro colonic fermentation. Supernatant will be used for metabolomics analysis (outcome 1) and selected fermentation time point pellets will be used for microbiota composition and functional analyses (outcome 3).

SECONDARY OUTCOMES:
Food intake using food diaries | 8 weeks
  Food diaries 3 times a week.
Assessment of the Gastrointestinal Symptom rating scale (GSRS) during the study | 8 weeks
  The gastrointestinal symptoms will be assessed during the baseline and protein supplementation period. Difference in the frequency and severity of gastrointestinal symptoms during the study will be assessed (15 questions with a scale of 1-7, minimum value 1, maximum 7, higher score correspond to a worse outcome)
Assessment of the bowel movement using the Bristol scale diary | 8 weeks
  The bowel movement will be assessed during the baseline and protein supplementation period by the Bristol scale diary. In the diary they write down the type of stool based on the scale which shows 7 pictures of different forms of stool, from watery diarrhea to compact. Participants are asked to choose the form of stool they have every day during the study.
Assessment of physical activity level | 8 weeks
  To assess the maintenance or difference of physical activity level during the baseline and dietary intervention by the AKTIVITETSVANOR questionnaire (Swedish questionnaire to assess physical activity frequency for 7 days).
Assessment of height | 4 weeks
  The height will be assessed in meters.
Assessment of body weight during the study | 4 weeks
  Participants will be weighted in order to have information of their body weight changes in kilograms during the study.
Assessment of body composition | 4 weeks
  Participants will be have their body composition measured using Tanita® full body scale. The obtained results by Tanita are: weight (kg), muscle mass (%) and kg), body water content (% and kg), fat mass (% and kg), basal energy expenditure (kcal and kJ) and BMI in kg/m^2.
Concentrations of faecal calprotectin | 4 weeks
  Difference in faecal levels of calprotectin during the study intervention
Fasting blood glucose level | 4 weeks
  Measurement of glucose in blood samples
Fasting blood insulin level | 4 weeks
  Measurement of insulin in blood samples
Fasting blood C-reactive protein level | 4 weeks
  Measurement of C-reactive protein in blood samples
Fasting blood cholesterol (total, LDL, and HDL) level | 4 weeks
  Measurement of cholesterol (total, LDL, and HDL) in blood samples (fasting state)
Fasting blood triglycerides level | 4 weeks
  Measurement of triglycerides in blood samples (fasting state)
Concentration of glucose - dietary challenge | 4 weeks
  Measurement of glucose in blood samples after the dietary challenge to check its level, compare with the fastening state and evaluate the area under the curve.
Concentration of insulin - dietary challenge | 4 weeks
  Measurement of insulin in blood samples after the dietary challenge to check its level, compare with the fastening state and evaluate the area under the curve.
Profile/composition of the gut microbiota after the intervention | 2 weeks
  Difference in the gut microbiota profile/composition 1 and 2 after the protein supplementation will be assessed by 16s/NGS. Alpha and Beta diversity will be measured and compared throughout these 2 weeks after the intervention. In the case of NGS, the genome sequence will be annotated and the resulting set of genes encoding for metabolic enzymes will be extracted. Data from shotgun metagenomics and metabolomics will be integrated by constructing dependency networks, with a special attempt to infer causal relationships among different variables.
Changes in the faecal metabolites using targeted and untargeted metabolomics after the intervention | 2 weeks
  Difference in faecal metabolites levels after the intervention will be measured. Targeted and untargeted metabolomics measurements will be used (e.g., short-chain fatty acids and branched chain fatty acids analyses, and polar and non polar metabolomics). Faecal samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared after 1 and 2 weeks of taking the protein supplements.
Breath test | 4 weeks
  From the subset of the participants, a breath sample will be collected by having them breathe into a breath sample collecting device (ReCIVA, Owlstone, UK), in order to measure volatile organic compounds by thermal desorption-gas chromatography coupled to ultra-resolution mass spectrometry (TD-GC-HRMS-Orbitrap).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Campus USÖ, Örebro University, Örebro, Sweden